CLINICAL TRIAL: NCT02003248
Title: A Feasibility Study to Evaluate Safety and Initial Effectiveness of ExAblate Transcranial MR Guided Focused Ultrasound for Unilateral Pallidotomy in the Treatment of Dyskinesia of Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2013-0051
Record Dates: First submitted 2013-12-01; First posted 2013-12-06 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Levodopa Induced Dyskinesia in Patients With Parkinson's Disease
Keywords: Parkinson's disease; ultrasound; dyskinesia; magnetic resonance
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dyskinesia of PD (Experimental): The proposed study is to evaluate the safety and initial effectiveness of the ExAblate Transcranial MRI-guided focused ultrasound (MRgFUS) treatment of patients with dyskinesia of Parkinson's Disease (PD)
  Interventions: Device: transcranial magnetic resonance guided focused ultrasound pallidotomy

INTERVENTIONS:
Device: transcranial magnetic resonance guided focused ultrasound pallidotomy — Focused ultrasound is an attractive method for non-invasive thermal ablation of soft tissue, including functional brain targets. Treatment begins by acquiring a series of MR images of the target organ. The physician then identifies a target volume in the MR images, and delineates the treatment contours on the images. Therapy planning software calculates the parameters required to effectively treat the defined target volume. During the treatment, an ultrasound transducer generates a point of focused ultrasound energy, called a sonication. The sonication raises the tissue temperature within a well-defined region, enabling neurophysiological assessment in the low range, and thermal coagulation at higher ranges. MR images acquired during sonication provide a quantitative, real-time temperature map of the target area to confirm the location of the sonication and the size of the affected region.

SUMMARY:
The proposed study is to evaluate the safety and initial effectiveness of the ExAblate Transcranial MRI-guided focused ultrasound (MRgFUS) treatment of patients with dyskinesia of Parkinson's Disease (PD)

* Safety: To evaluate the incidence and severity of adverse events (AE/AEs) associated with ExAblate Transcranial MRgFUS treatment of dyskinesia of PD
* Effectiveness: To determine the level of effectiveness of the ExAblate Transcranial MRgFUS treatment of dyskinesia of PD.Efficacy will be determined utilizing the UPDRS-IV for dyskinesia in PD from examinations at baseline and every 3-Months post-ExAblate treatment.

This study is designed as a prospective, single-site, single arm, nonrandomized study. Assessments will be made before and three months after MRgFUS for clinical symptom relief, quality of life (QoL) improvements, and safety of MRgFUS in the treatment of LID. Relative Safety will be evaluated using a common description of Significant Clinical Complications for patients treated in this study. This study will be performed on the 3T MR scanners.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between 20 and 80 years, inclusive
* Willing to give consent and able to attend all study visits
* Diagnosis of PD as confirmed from clinical history and examination by a movement disorder neurologist
* Show unequivocal response to dopaminergic agents, specified as at least 33% improvement in United Parkinson Disease Rating Scale motor subscore (UPDRS-III) and diagnosed as idiopathic PD for more than 5 years.
* GPi nucleus of pallidum can be targeted by the ExAblate device. The GPi region of the pallidum must be apparent on MRI such that targeting can be performed with either direct visualization or by measurement from a line connecting the anterior and posterior commissures of the brain.
* Able to communicate sensations during the ExAblate MRgFUS treatment
* One of dyskinesia rating scores greater than or equal to 2 in UPDRS-IV A-32, 33, & 33.
* Stable doses of all medications for 30 days prior to study entry and for the duration of the study.
* Inclusion and exclusion criteria have been agreed upon by two members of the medical team.

Exclusion Criteria:

* Unstable cardiac status including: Unstable angina pectoris on medication / Patients with documented myocardial infarction within six months of protocol entry / Congestive heart failure requiring medication (other than diuretic) / Patients on anti-arrhythmic drugs
* Exhibit any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within a 12 month period: Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household). / Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use) / Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct) / Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
* Severe hypertension (diastolic BP > 100 on medication)
* Contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
* Severely impaired renal function (estimated glomerular filtration rate < 45ml/min/1.73 m2) or receiving dialysis
* History of abnormal bleeding and/or coagulopathy
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
* Active or suspected acute or chronic uncontrolled infection
* History of intracranial hemorrhage
* Cerebrovascular disease (multiple CVA or CVA within 6 months)
* Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time.)
* Symptoms and signs of increased intracranial pressure (e.g. headache, nausea, vomiting, lethargy, and papilledema)
* Are participating or have participated in another clinical trial in the last 30 days
* Unable to communicate with the investigator and staff.
* Presence of any other neurodegenerative disease like parkinson-plus syndromes suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease.
* Anyone suspected to have the diagnosis of idiopathic Parkinson's disease. This includes excluding anyone with the presence of parkinsonian features including bradykinesia rigidity, or postural instability.
* Presence of significant cognitive impairment as determined with a score ≤ 24 on the Mini Mental Status Examination (MMSE)
* History of immunocompromise, including patient who is HIV positive
* Known life-threatening systemic disease
* Patients with a history of seizures within the past year
* Patients with current or a prior history of any psychiatric illness will be excluded. Any presence or history of psychosis will be excluded. Patients with mood disorders including depression will be excluded. For the purpose of this study, we consider a significant mood disorder to include any patient who has: been under the care of a psychiatrist for over 3 months / taken antidepressant medications for greater than 6 months / has participated in cognitive-behavioral therapy / been hospitalized for the treatment of a psychiatric illness / received transcranial magnetic stimulation / received electroconvulsive therapy
* Patients with risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter, PT > 14, PTT > 36 or INR > 1.3) or a documented coagulopathy
* Patients with brain tumors
* Any illness that in the investigator's opinion preclude participation in this study.
* Pregnancy or lactation.
* Legal incapacity or limited legal capacity.
* Patients who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia
* Prior intracranial surgery
* Calcifications in the sonication pathway that cannot be avoided by tailoring the treatment plan
* More than 20% of the scalp in the sonication pathway is covered by scars, scalp disorders (e.g., eczema) or atrophy of the scalp
* Clips or other metallic implanted objects in the sonication pathway, except shunts.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11-08 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
the unified dyskinesia rating scale (UdysRS) and UPDRS part IV | 3 months after treatment
  Dyskinesia will be assessed for each treated PD patient using the UDysRS and UPDRS part IV at baseline before treatment and at post-treatment intervals: 1 week, 1 month, and 3 months, 6 months and 12 months. The validated rating assessment of dyskinesia will be administered by a movement disorder neurologist or physical therapy specialist in an outpatient clinic setting. The primary measure utilized in this protocol will be a reduction in the contralateral upper extremity. Additionally, a total/overall dyskinesia score will be obtained for each patient at each time interval by summing the appendicular and axial scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Jung NY, Park CK, Kim M, Lee PH, Sohn YH, Chang JW. The efficacy and limits of magnetic resonance-guided focused ultrasound pallidotomy for Parkinson's disease: a Phase I clinical trial. J Neurosurg. 2018 Aug 10;130(6):1853-1861. doi: 10.3171/2018.2.JNS172514. Print 2019 Jun 1. PMID 30095337